CLINICAL TRIAL: NCT05550948
Title: Use of Transcranial Photobiomodulation to Improve Cognition and Self-Reported Outcomes in Survivors of Childhood Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Device Feasibility
Other Study IDs: PBMP; NCI-2022-09116 (Other: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: ALL; Hodgkin Lymphoma; Cancer; Survivorship
MeSH Terms: conditions — Hodgkin Disease; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The proposed study is a double-blind, randomized placebo-controlled pilot study of remotely delivered tPBM paired with cognitive training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- alpha tPBM + cognitive training (Experimental): three days per week for a 2-month intervention period (5 ALL and 5 HL)
  Interventions: Device: Transcranial photobiomodulation (tPBM) - Mobile System
- gamma tPBM + cognitive training (Experimental): three days per week for a 2-month intervention period (5 ALL and 5 HL)
  Interventions: Device: Transcranial photobiomodulation (tPBM) - Mobile System
- sham tPBM + cognitive training (Experimental): Sham stimulations will act as the control for this study three days per week for a 2-month intervention period (5 ALL and 5 HL)
  Interventions: Device: Transcranial photobiomodulation (tPBM) - Mobile System

INTERVENTIONS:
Device: Transcranial photobiomodulation (tPBM) - Mobile System — The Vielight NeURO device delivers 810 nm near infrared light via four (4) transcranial LED modules. The LED modules target brain regions associated with a variety of cognitive functions. It can deliver light at two frequencies: Alpha (10 Hz) and Gamma (40 Hz). Alpha oscillations are prominent in healthy brains during wakeful resting and gamma oscillations are associated with activities associated with focus, memory, and cognition.
  Other Names: Vielight portable tPBM NeURO device.

SUMMARY:
Survivors of childhood cancer are at greater risk for long-term cognitive impairments that include attention, executive function, intelligence, memory, and processing speed. The participants are a survivor of acute lymphoblastic leukemia (ALL) or Hodgkin's lymphoma (HL). Because of your treatment the participant may have developed trouble with thinking and learning.

Primary Objective

To evaluate the feasibility of using home-based tPBM paired with remote cognitive training to improve cognitive performance in survivors of ALL and HL.

Secondary Objectives

To estimate the potential efficacy of alpha and gamma frequency tPBM on cognitive performance in survivors of ALL and HL.

Exploratory Objectives

To estimate the effects of home-based tPBM paired with remote cognitive training on patient reported symptoms of executive dysfunction, sleep, depression, anxiety, fatigue, and pain in survivors of ALL and HL.

DETAILED DESCRIPTION:
Survivors with ALL and HL with identified executive function impairment will be randomized to receive stimulation with alpha tPBM + cognitive training, gamma tPBM + cognitive training or sham tPBM + cognitive training three days per week for a 2-month intervention period The tPBM will be applied to nodes in the default mode network.

ELIGIBILITY:
Inclusion Criteria:

* Completed treatment for acute lymphoblastic leukemia (ALL) or Hodgkin's Lymphoma (HL) at SJCRH.
* Enrolled in SJLIFE, and less than 21 years of age at diagnosis.
* 18 years of age or older at time of enrollment.
* 2 years or greater post-treatment completion of cancer directed therapy and not currently receiving any cancer directed therapy.
* English language proficiency.
* Access to WiFi.
* Executive dysfunction defined as having an age-adjusted standard score less than 16th percentile on objectively assessed cognitive test or patient-reported executive dysfunction defined as having a standard score greater than 84th percentile within 3 years of time of enrollment.

Exclusion Criteria:

* Estimated intelligence score less than 80.
* Currently taking medication intended to treat neurocognitive impairment (i.e., stimulants).
* Major psychiatric condition.
* Alcohol abuse in the past year (AUDIT) [greater than or equal to 13 for women and greater than or equal to 15 for men]. The Alcohol Use Disorders Identification Test (AUDIT) will be used to screen for individuals who have active alcohol-use disorders.
* Drug abuse in the past year (DAST-10) [ greater than or equal to 3 for women or men] The Drug Abuse Screen Test (DAST-10) will be used to screen for individuals with active drug abuse.
* History of neurologic condition or genetic disorder associated with neurocognitive impairment unrelated to cancer diagnosis or treatment.
* Enrolled on another independent cognitive intervention protocol within the last year.
* Female participants who are pregnant or lactating (determined by participant self-report due to the remote nature of this study)
* Tattoo or artificial marking in the area where the device will be positioned.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants who completed a two-month trial of paired photobiomodulation (PBM) therapy and cognitive training | 4 months after participant enrollment
  The trial will be considered feasible if at least 15 of 30 survivors are able to complete 18 of 24 sessions (PBM along with cognitive training).

SECONDARY OUTCOMES:
CNS Vital Signs adaptions of the Rey auditory verbal learning test (RVLT). | 2 month and 4 months after enrollment
  RVLT is a test that evaluate working memory.
CNS Vital Signs adaptions of the Rey visual design learning (RVDL) test. | 2 month and 4 months after enrollment
  RVDL is a test that evaluate working memory.
CNS Vital Signs implemented Stroop color and word test. | 2 month and 4 months after enrollment
  The Stroop test is a test that evaluates Inhibitory control.
CNS Vital Signs implemented Shifting Attention Test. | 2 month and 4 months after enrollment
  The Shifting attention test and Stroop test are tests that are used to measure cognitive flexibility.
CNS Vital Signs implementation of the Continuous Performance Test (CPT). | 2 month and 4 months after enrollment
  The CPT test is a test that evaluates attention.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Phillips, MD,PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols